CLINICAL TRIAL: NCT06396598
Title: SyMPLER: Patient- and Caregiver-Triggered Palliative Referrals Via an Electronic Symptom Monitoring Program
Brief Title: Electronic Symptom Monitoring Program for Triggered Palliative Referrals in Patients With Thoracic Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Julia Agne, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-23149; NCI-2024-00269 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-04-12; First posted 2024-05-02 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Malignant Thoracic Neoplasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (electronic symptom monitoring program) (Experimental): Patients and their caregivers participate use the electronic symptom monitoring program to log symptoms QW for 24 weeks. Patients and their caregivers also watch a video and review education materials prior to starting the remote symptom monitoring program.
  Interventions: Other: Educational Activity; Other: Electronic Health Record Review; Other: Internet-Based Intervention; Other: Media Intervention; Other: Survey Administration

INTERVENTIONS:
Other: Educational Activity — Review education materials
Other: Electronic Health Record Review — Ancillary studies
Other: Internet-Based Intervention — Participate use the electronic symptom monitoring program to log symptoms
Other: Media Intervention — Watch a video
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates earlier symptom management through remote electronic symptom monitoring (such as through an app on patient's phone), and accessibility of palliative care self-referral by patients with thoracic cancer and caregivers by proxy (legal representative). Thoracic cancer occurs in the chest and often causes symptoms for patients. Patients and/or their caregivers are often unable to attend in-person clinic visits for various reasons. The most frequently reported symptom by patients at initial palliative care consultations is pain, and caregivers' most common concerns are pain management for the patient, stress reduction, and fears about patient decline. Earlier palliative care referral can help control these symptoms before they worsen, providing a better quality of life for patients and caregivers. improve physical and emotional functioning for patients and caregivers in cancer care. This study may help researchers learn how an electronic symptom monitoring program may provide an earlier and more accessible way for patients with thoracic cancer to receive palliative care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Develop and assess feasibility of a remote electronic symptom monitoring program with a prompted option for palliative care self-referral for patients or caregivers by proxy after diagnosis of a thoracic malignancy.

SECONDARY OBJECTIVE:

I. Evaluate palliative care referral patterns after implementation of a remote electronic symptom monitoring program.

OUTLINE:

Patients and their caregivers use the electronic symptom monitoring program to log symptoms once a week (QW) for 24 weeks. Patients and their caregivers also watch a video and review education materials prior to starting the remote symptom monitoring program.

After completion of study intervention, participants are followed up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS: Age ≥ 18 years
* PATIENTS: Diagnosed with any stage (1-4) or type (non-small cell lung cancer, small cell lung cancer, mesothelioma, thymic carcinoma) of thoracic malignancy
* PATIENTS: ≥ 2 visits at the Ohio State University Comprehensive Cancer Center (OSUCCC) Thoracic Oncology Clinic
* PATIENTS: Study enrollment within 12 weeks of initial Thoracic Medical Oncology appointment
* PATIENTS: Ability to understand and willingness to sign an informed consent document (or indicate approval or disapproval by another means)
* PATIENTS: Ability to read and understand English
* PATIENTS: Access to a device with email or text messaging capability
* CAREGIVERS: Age ≥ 18 years
* CAREGIVERS: Identified by patient participant as primary caregiver
* CAREGIVERS: Corresponding patient participant has consented to participate in the study
* CAREGIVERS: Ability to understand and willingness to sign an informed consent document (or indicate approval or disapproval by another means)
* CAREGIVERS: Ability to read and understand English
* CAREGIVERS: Access to a device with email or text messaging capability

Exclusion Criteria:

* PATIENTS: Patients who have been previously referred to ambulatory palliative care are excluded from participation
* PATIENTS: Prisoners are excluded from participation
* PATIENTS: Pregnant patients are excluded from participation
* PATIENTS: Patients who lack capacity for medical decision-making as determined by their primary oncologist are excluded from participation
* PATIENTS: There is NO exclusion criteria pertaining to Eastern Cooperative Oncology Group (ECOG) performance status, laboratory values, prior cancer diagnoses, presence of comorbidities or brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Frequency of symptom logging | At 6 months after enrollment
  Will estimate that ≥ 50% of patient participants will log symptoms at least monthly through the remote electronic symptom monitoring program.
Proportion of patients enrolled (Feasibility) | At enrollment and 3 months
  Descriptive statistics will include study enrollment rates (eligible vs. ineligible participants, consented vs. refused), completion rate of weekly symptom monitoring (patient vs. caregiver by proxy), and person requesting palliative care services (patient vs. caregiver by proxy vs. medical provider), if applicable. Will be considered feasible if within 20% of target enrollment.
Symptom scores and Palliative Referral Association | At enrollment and 3 months and 6 months
  Symptom scores (Edmonton Symptom Assessment Scale revised with Constipation and Sleep [ESAS-r-CS]) reported by patients and caregivers will be tracked and their association with palliative care referral, if applicable, will be assessed.
Patient and Caregiver Symptom Reporting Congruency | At enrollment and 3 months and 6 months
  Descriptive statistics will be used to assess for congruency between patient and proxy-reported symptom assessments. Patients' oncologic treatment (chemotherapy, immunotherapy, radiation therapy, surgery) will be abstracted from the electronic medical record (EMR) at the time of each ESAS-r-CS survey completed by either the patient or caregiver by proxy.

SECONDARY OUTCOMES:
Palliative care referral patterns | Up to 24 months
  Palliative care referrals pre- and post- launch of the SyMPLER study will be evaluated for trends. Historical control data collecting palliative referrals by month will be compared between groups (pre-post- launch).

CONTACTS AND LOCATIONS:
Overall Officials: Julia L Agne, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu